CLINICAL TRIAL: NCT00284076
Title: L-Arginine in the Treatment of Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 357; T32HL007708 (NIH); P50HL083800 (NIH); P01AI050153 (NIH); R01HL075774 (NIH); R01HL063685 (NIH)
Record Dates: First submitted 2006-01-27; First posted 2006-01-31 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Diseases; Peripheral Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Vascular Diseases | interventions — Arginine

INTERVENTIONS:
Drug: L-arginine

SUMMARY:
To assess the effects of L-arginine upon functional status (treadmill exercise testing; quality of life) and limb blood (by mercury strain gauge plethysmography) in peripheral arterial disease.

DETAILED DESCRIPTION:
BACKGROUND:

Peripheral arterial disease is a common disorder effecting up to 15% of men over age 55 and women over age 65. Patients with peripheral arterial disease are at increased risk for stroke, myocardial infarction or other adverse vascular outcomes. Therapy for this disorder is currently limited with only 2 FDA approved drugs (Pentoxifylline, cilostazol). These agents improve walking distance by 10 to 40 percent. Other agents such as verapamil and prostacyclin analogs have significant side effects. Although therapy with angiogenesis inducers, including injections of plasmid constructs for vascular endothelial growth factor (VEGF) or VEGF protein, is beneficial, the widespread applicability of this therapy is questionable. The study used an alternative approach, which may be safer and more effective. The basis for this approach is the ability of L-arginine to enhance endogenous vascular nitric oxide production, improving blood flow acutely. Furthermore, since several angiogenic growth factors may act at least partially through the production of nitric oxide, this therapy could produce a sustained benefit by the induction of an increase in skeletal muscle capillary density.

DESIGN NARRATIVE:

A randomized placebo-controlled trial to assess the effects of L-arginine on functional status was performed in patients with peripheral arterial disease. Blood flow was assessed by Doppler and plethysmography and measures of nitric oxide synthesis (plasma and urinary nitrogen oxides) were performed. The effect of L-arginine on treadmill walking distance was determined. The potential for L-arginine induced angiogenesis was assessed using magnetic resonance angiography.

There were two separate studies of oral L-arginine. The first was a dose ranging study involving 80 patients receiving four different doses of L-arginine (9 grams, 6 grams, 3 grams, or 0 grams). The dosing of L-arginine was performed in a randomized placebo-controlled fashion. Patients receive six weeks of therapy. Patients with diabetic retinopathy, active malignancy or previous malignancy in a state of remission, or autoimmune disorders were excluded. Ophthalmological exams were performed to screen for pathological angiogenesis in the retina. After the completion of the dose response study, the investigators studied the safety and efficacy of prolonged (12 months) L-arginine therapy. The primary end point was absolute claudication distance (ACD) and a statistical analysis was performed of the logarithm ACDT / ACDB. A treadmill was performed at one month after cessation of therapy to determine if there was a structural alteration of the indices of limb hemodynamics including the ankle brachial index (ABI) and plethysmography was performed at 6 and 12 months of therapy and at 1 month after sensation of therapy. The study correlated measures of limb blood flow with evidence of increased nitric oxide synthesis by measuring urinary nitrogen oxide. Flow mediated vasodilation (FMVD) of the brachial artery was measured. The choice of monitoring flow mediated vasodilation of the brachial artery, while appropriate for showing a systemic enhancement of nitric oxide synthesis, would not directly support an improvement of endothelial function in the vascular bed of interest.

Asymmetric dimethylarginine (ADMA) was measured with the prediction that patients with elevated ADMA levels, depressed urinary nitrogen oxides and reduced FMVD might be more responsive to L-arginine therapy. A second aim of the protocol was to determine if the chronic enhancement of nitric oxide synthesis by L-arginine supplementation had an enduring effect on conduit vessel structure. The ankle brachial index, plethysmography, and MR perfusion imaging were performed at 0, 6 and 12 months on therapy, and at 1 month after cessation of therapy.

ELIGIBILITY:
Patients with diabetic retinopathy, active malignancy or previous malignancy in a state of remission, or autoimmune disorders will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Cooke — Stanford University

REFERENCES:
- [Derived] Wilson AM, Shin DS, Weatherby C, Harada RK, Ng MK, Nair N, Kielstein J, Cooke JP. Asymmetric dimethylarginine correlates with measures of disease severity, major adverse cardiovascular events and all-cause mortality in patients with peripheral arterial disease. Vasc Med. 2010 Aug;15(4):267-74. doi: 10.1177/1358863X10364552. Epub 2010 May 19. PMID 20484311